CLINICAL TRIAL: NCT05667636
Title: Early Salvage Stereotactic Radiotherapy (esSBRT) for Biochemical Failure After Radical Prostatectomy :a Phase II Study
Brief Title: Early Salvage Stereotactic Radiotherapy for Biochemical Failure After RP
Acronym: esSBRT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: Alessia Farneti (Unknown); Adriana Faiella (Unknown); Marta Bottero (Unknown); Pasqualina D'Urso (Unknown); Valeria Landoni (Unknown); Antonella Soriani (Unknown); Luca Bertini (Unknown)
Responsible Party: Principal Investigator, Giuseppe Sanguineti, Professor, Regina Elena Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RS1705/22 (2678)
Record Dates: First submitted 2022-09-30; First posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Prostatic Neoplasm
Keywords: prostate cancer;; biochemical recurrence;; salvage radiotherapy;; SBRT;
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single arm, non randomized (Experimental): SBRT 30 Gy/ 5 fractions
  Interventions: Radiation: salvage SBRT
- radiation, SBRT (Experimental): SBRT 30 Gy/5 fractions to the prostatic bed +/- 25 Gy/5 fractions to the pelvic lymphnodes
  Interventions: Radiation: salvage SBRT

INTERVENTIONS:
Radiation: salvage SBRT — steretactic body radiation therapy in the setting of salvage radiotherapy for prostate cancer

SUMMARY:
After radical prostatectomy, 30-60% of patients will develop recurrent disease. Salvage radiotherapy, usually at 2 Gy per fraction, is the main treatment option for these patients.

The aim of the present study is to determine the 3-yr biochemical failure free survival of the stereotactic approach in 5 fractions in the context of salvage radiotherapy for biochemical failure after radical prostatectomy.

DETAILED DESCRIPTION:
The present study aims at delivering 30 Gy to the prostatic bed in 5 fractions. At the same time, the pelvic nodes will be covered to 25 Gy, but in those patients considered at low risk of nodal involvement. In patients with evidence of macroscopic disease at the tumor bed through DCE-MRI, 40 Gy will be delivered in 5 fractions.

Selected patients will receive 6-month LHRH analogue preceded by Bicalutamide tablet 50 mg, daily, for 2 weeks to control for possible tumor flare.

ELIGIBILITY:
Inclusion Criteria:

* - Able and willing to provide informed consent;
* Pathologically proven diagnosis of prostatic adenocarcinoma;
* Biochemical failure (2 consecutive PSA rises above 0.2 ng/ml) after radical prostatectomy;
* No regional or distant metastases;
* Eastern Cooperative Oncology Group performance status 0-1

Exclusion Criteria:

* - Previous local treatment of the prostate with radiotherapy, brachytherapy, cryosurgery, high-intensity focused ultrasound or cryotherapy;
* Previous radiotherapy to the pelvis;
* Previous or current symptomatic vesicourethral anastomotic stenosis post-RP (weak stream, straining to void, hesitancy and incomplete bladder emptying);
* PSA level at sRT> 2 ng/ml;
* (Each single) Lesion volume within the prostatic fossa at mpMR >5 cc;
* Previous chemotherapy for malignancy in past 5 years;
* Previous androgen deprivation for biochemical failure after RP;
* Contraindication to short term AD (in case of Px)
* Presence of nodal or distant metastasis, as confirmed by magnetic resonance (MR) or PET/CT
* Pathologically positive lymph nodes (pN+) at RP;
* Serious medical comorbidities or other contraindications to radiotherapy
* Presence of active inflammatory bowel disease;
* Presence of active connective tissue disease;
* Unable or unwilling to complete quality of life questionnaires

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 103 (Estimated)
Dates: Start 2022-09-27 (Actual); Primary Completion 2023-09-27 (Estimated); Study Completion 2024-09-27 (Estimated)

PRIMARY OUTCOMES:
3-yr BFFS | 3-years
  The primary objective of the study is 3-yr biochemical failure free survival of the stereotactic approach in 5 fractions in the context of salvage radiotherapy for biochemical failure after RP

SECONDARY OUTCOMES:
3-y OS | 3-years
  The secondary objective is 3-yr overal survival
3-y LC | 3-years
  The secondary objective is 3-yr locoregional control assessed with PSA
3-y MFS | 3-years
  The secondary objective is 3-yr metastases free survival
3-y GU GI tox | 3-years
  The secondary objective is 3-yr genitourinary and gastrointestinal toxicity according to CTCAE v5.0
3-y QoL | 3-years
  The secondary objective is 3-yr quality of life (FACT-P, IIF-5, ICIQ-SF, IPSS, IBQD)
3-y - Patient satisfaction with treatment | 3-years
  The secondary objective is 3-y patient satisfaction with treatment (FACIT-TS-G)

CONTACTS AND LOCATIONS:
Locations (1):
- Regina Elena National Cancer Institute, Rome, Italy

IPD SHARING:
Plan to Share IPD: No